CLINICAL TRIAL: NCT02318459
Title: High Intensity Interval Training for thE Rehabilitation of Geriatric Patients - a Feasibility Pilot studY.
Brief Title: High Intensity Interval Training in Geriatrics
Acronym: HIITERGY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jean-Luc Reny, Head of division, Internal medicine and rehabilitation Trois-Chêne, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 13-257
Record Dates: First submitted 2014-11-07; First posted 2014-12-17 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Muscle Weakness; Gait, Unsteady
MeSH Terms: conditions — Muscle Weakness; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high intensity interval training-HIIT (Experimental): HIIT 4 times a week, 30 minutes duration
  Interventions: Other: high intensity interval training-HIIT
- Traditionnal rehabilitation (Active Comparator): Traditionnal group rehabilitation 3 times a week, 1 hour duration.
  Interventions: Other: Traditionnal group rehabilitation

INTERVENTIONS:
Other: high intensity interval training-HIIT — HIIT 4 times a week, 30 minutes duration
  Arms: high intensity interval training-HIIT
Other: Traditionnal group rehabilitation — Traditionnal group rehabilitation, 3 times a week, 1 hour duration
  Arms: Traditionnal rehabilitation

SUMMARY:
This is a pilot study for evaluating the feasibility of using High Intensity Interval Training in geriatric hospitalized patients compared to the standard current rehabilitation practice.

DETAILED DESCRIPTION:
High Intensity Interval Training (HIIT) has shown a superior effectiveness and efficiency when compared to Moderate Intensity Continuous Training (MICT) in several types of patients and in healthy subjects. There are no data on HIIT in a general geriatric population. This study is a pilot study evaluating the feasibility of using HIIT in geriatric hospitalized patients compared to the standard current rehabilitation practice without HIIT. It is our desire to perform a larger randomized comparative trial between HIIT and MICT if the pilot study proves its feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older hospitalized for rehabilitation after an acute medical condition
* Expected duration of the rehabilitation ≥ 2 weeks
* Ability to follow instructions to perform a Timed up and Go Test
* Ability to perform exercises
* Willing to participate in 4 sessions of HIIT per week for 2 weeks

Exclusion Criteria:

* Any acute condition with tachycardia, hypotension or fever.
* Abnormal cycle ergometer stress test with
* significant ECG modification
* decrease of more than 20 mmHg of the blood pressure with exercise
* angina
* ST depression at a workload <6 METs
* Inability to reach an intensity of 15/20 in the Borg's scale of perceived exertion
* Any unresolved acute medical or surgical condition of the following kind:
* acute heart failure
* acute coronary syndrome < 1 month
* strole < 1 month
* active pericarditis / myocarditis / endocarditis
* thromboembolic disease with < 2 weeks of anticoagulation
* acute infection requiring intravenous treatment
* ongoing intravenous perfusion
* surgery < 2 months
* recent bone fracture
* Previous episode of primary cardiac arrest (ie, cardiac arrest that did not occur in the presence of an acute myocardial infarction or during a cardiac procedure).
* Severe heart failure (NYHA III and IV)
* Severe stenotic or regurgitant valvular disease
* Uncontrolled hypertension at rest (SBP≥160mmHg, DBP≥100mmHg)
* Uncontrolled dysrhythmia
* Non-sustained ventricular tachycardia with exercise
* Implanted defibrillator
* Obstructive cardiomyopathy
* Resting HR > 100/min
* Severe peripheral artery disease
* Severe COPD (VEMS < 50%)
* Exercise-induced asthma
* Oxygen dependency
* Muscular-skeletal anomaly that may limit exercise participation
* Delirium
* Inability to follow instructions
* Inability to consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who complete the rehabilitation program | 2 weeks

SECONDARY OUTCOMES:
Distance walked in the 6MWT | 2 weeks
Muscle strength assessed for the upper and lower extremities | 2 weeks
  upper extremity : handgrip strength using the Baseline Pneumatic Bulb Hand Dynamometer Pinch Gauge; Lower exremity : knee flexion & extension and ankle flexion & extension using Microfet2™portable Dynamometer.
Step variability changes as a measure of quality of ambulation | 2 weeks
  Variability measured with GaitRite step analysis system

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Reny, MD, PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpital des Trois-Chêne (HUG), Geneva, Thônex, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pires Peixoto R, Trombert V, Poncet A, Kizlik J, Gold G, Ehret G, Trombetti A, Reny JL. Feasibility and safety of high-intensity interval training for the rehabilitation of geriatric inpatients (HIITERGY) a pilot randomized study. BMC Geriatr. 2020 Jun 5;20(1):197. doi: 10.1186/s12877-020-01596-7. PMID 32503465